CLINICAL TRIAL: NCT00935220
Title: An Open Label, Phase I Trial to Investigate the Pharmacokinetics and Pharmacodynamics of Linagliptin (BI 1356) 5 mg After Single and Multiple Oral Administration in Patients With Type 2 Diabetes Mellitus of African American Origin for 7 Days
Brief Title: Pharmacokinetics and Pharmacodynamics Trial With Linagliptin (BI 1356) 5mg in African American Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1218.55
Record Dates: First submitted 2009-07-01; First posted 2009-07-08 (Estimated); Results first posted 2011-11-10 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — WW Domain-Containing Oxidoreductase

ARMS (1):
- linagliptin (Experimental): Pharmacokinetic (PK)/Pharmacodynamic (PD) investigation
  Interventions: Drug: linagliptin QD (once daily) for 7 days

INTERVENTIONS:
Drug: linagliptin QD (once daily) for 7 days — dipeptidyl peptidase IV (DPP-4) activity will be measured as PD response to drug administration

SUMMARY:
The objective of this trial is to investigate the pharmacokinetics and pharmacodynamics of linagliptin (BI 1356) 5 mg administered orally in patients with Type 2 diabetes mellitus of African American origin.

ELIGIBILITY:
Inclusion criteria:

1. Glycosylated haemoglobin >=7 and <= 10%
2. Age >=21 and <= 65
3. Body Mass Index >=18.5 and <=38 kg/m2
4. African American origin
5. Signed and dated informed consent prior to admission to the study

Exclusion criteria:

1. Any finding of the medical examination considered clinically relevant by the Investigator
2. Clinically relevant concomitant diseases like renal insufficiency, cardiac insufficiency New York Heart Association (NYHA) II-IV, known cardiovascular disease including hypertension >160-100 mmHg (under current treatment), stroke and transient ischemic attack (TIA).
3. Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders besides type 2 diabetes
4. Clinically relevant diseases of central nervous system or psychiatric disorders or relevant neurological disorders besides polyneuropathy
5. Diagnosis of sickle cell anemia or known chronic anemia
6. History of chronic or relevant infections (for example human immunodeficieny virus (HIV), Hepatitis B)
7. History of relevant allergy/hypersensitivity
8. Intake of drugs with a long half life (>24hours) within at least one month or less than 10 half lives of the respective drug prior to administration except allowed co medication
9. Alcohol abuse, drug abuse
10. Any laboratory value of clinical relevance that is outside an acceptable range
11. Change of drug dosing of allowed co medication
12. Any (electrocardiogram) ECG value outside the reference range and of clinical relevance.
13. Fasted glucose >270 mg/dl or randomly determined blood glucose >400 mg/dl on two consecutive days during screening or wash out
14. Serum creatinine above upper limit normal at screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- United States (6):
  - 1218.55.0006 Boehringer Ingelheim Investigational Site, Cypress, California
  - 1218.55.0008 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1218.55.0004 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.55.0005 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1218.55.0003 Boehringer Ingelheim Investigational Site, New York, New York
  - 1218.55.0001 Boehringer Ingelheim Investigational Site, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Linagliptin 5mg: Linagliptin 5mg once daily
Period: Overall Study
Arm/Group | Linagliptin 5mg
Started | 41
Completed | 39
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Other reason (not specified) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black / African American | 41
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 30.93 (3.90)

OUTCOME MEASURES:

1. Secondary Outcome: Treatment Emergent Adverse Events
Description: Frequency of patients with AEs
Time Frame: 21 days
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 41
Participants
  Patients with any adverse events (AEs) | 16
  Patients with severe AEs | 0
  Patients with drug-related AEs | 7
  Discontinuation due to AEs | 0

2. Secondary Outcome: Electrocardiogram (ECG), Vital Signs, Physical Finding or Laboratory Finding Abnormalities
Description: 12-lead-Electrocardiogram (ECG), vital sign (blood pressure and pulse rate), physical finding and laboratory abnormalities
Time Frame: 21 days
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 41
Participants
  ECG abnormalities | 0
  Vital signs abnormalities | 0
  Physical finding abnormalities | 0
  Laboratory finding abnormalities | 5

3. Primary Outcome: Linagliptin: AUC_τ,ss
Description: area under the concentration time curve (AUC_τ) of linagliptin in plasma at steady state over a uniform dosing interval
Time Frame: 24 hours
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 39
nmol*h/L | 194 (25.8)

4. Primary Outcome: Linagliptin: C_max,ss
Description: maximum concentration of linagliptin in plasma at steady state
Time Frame: 24 hours
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 39
nmol/L | 16.4 (40.9)

5. Secondary Outcome: Patients With Electrocardiogram (ECG), Vital Signs, Physical Finding or Laboratory Finding Abnormalities Reported as an Adverse Event
Description: Patients with Electrocardiogram (ECG), vital signs, physical finding reported as an adverse event
Time Frame: 21 days
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 41
Participants | 0

6. Secondary Outcome: Linagliptin: AUC_0-24
Description: area under the concentration time curve of linagliptin in plasma over the time interval from 0 to 24h after administration of the first dose
Time Frame: 24 hours
Population: Treated set- All patients with values for the area under the concentration time curve of the analyte in plasma over the time interval from 0 to 24 h after administration of the first dose (AUC_0-24) for Linagliptin
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 41
nmol*h/L | 137 (32.4)

7. Primary Outcome: DPP-4 Inhibition: E_24,ss
Description: Plasma DPP-4 inhibition at trough under steady state conditions. Plasma DPP-4 inhibition is derived by calculating (1-(activity in presence of linagliptin)/baseline activity))*100%, where 'activity' is the activity of the DPP-IV enzyme.
Time Frame: One single measurement 24 h after drug administration under steady state conditions
Population: Treated set
Measure: Median (Full Range); unit: Percent (of inhibition)
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 37
Percent (of inhibition) | 84.7 [72.2 to 91.9]

8. Secondary Outcome: Linagliptin: C_max
Description: maximum concentration of linagliptin in plasma on Day 1
Time Frame: 24h
Population: Treated set - All patients with values for the maximum measured concentration of linagliptin in plasma (C_max)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 41
nmol/L | 10.9 (57.6)

9. Secondary Outcome: DPP-4 Inhibition: E_24
Description: Plasma DPP-4 inhibition 24 hours after first dose. Plasma DPP-4 inhibition is derived by calculating (1-(activity in presence of linagliptin)/baseline activity))*100%, where 'activity' is the activity of the DPP-IV enzyme.
Time Frame: One single measurement 24 h after drug administration
Population: Treated set
Measure: Median (Full Range); unit: Percent (of inhibition)
Arm/Group | Linagliptin 5mg
Number analyzed (Participants) | 39
Percent (of inhibition) | 75.2 [52.0 to 89.8]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Linagliptin 5mg
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 5/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin 5mg (N=41)
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.